CLINICAL TRIAL: NCT01190176
Title: Gynaecological Follow-up of a Subset of HPV-015 Study Subjects
Brief Title: Gynaecological Follow-up of a Subset of HPV-015 (NCT00294047) Study Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113617; 2009-017282-35 (EudraCT Number)
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; HPV vaccine; Cervical neoplasia; Human papillomavirus; Papillomavirus; Cervical cancer; Human papillomavirus (HPV) type 16/18 infections
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- HPV-062 study subjects Group (Experimental): HPV-015 (NCT00294047) study subjects who had normal cervical cytology, but tested positive for oncogenic HPV infection at their concluding HPV-015 (NCT00294047) study visit or were pregnant, so that no cervical sample could be collected at their concluding HPV-015 (NCT00294047) study visit.
  Interventions: Procedure: Gynaecological follow-up; Biological: Cervarix; Biological: Placebo control

INTERVENTIONS:
Procedure: Gynaecological follow-up — Subjects will receive a gynaecological follow-up with cytology and oncogenic HPV DNA testing every 12 months, for up to a maximum of four years.
Biological: Cervarix — Subjects received 3 doses of the HPV vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule in the primary study HPV-015.
Biological: Placebo control — Subjects received 3 doses of the control [Al(OH)3] administered intramuscularly according to a 0, 1, 6 month vaccination schedule in the primary study HPV-015.

SUMMARY:
This study is intended to provide up to a maximum of four years of annual oncogenic human papillomavirus (HPV) DNA testing and cervical cytology examination for NCT00294047 study subjects who displayed normal cervical cytology but tested positive for oncogenic HPV infection at their concluding NCT00294047 study visit.

Women who were pregnant at their concluding NCT00294047 study visit may also be included in this study, as no cervical sample could be collected at that visit.

The objectives and outcome measures of the primary phase (NCT00294047) are presented in a separate protocol posting.

DETAILED DESCRIPTION:
Cervarix or Control [Al(OH)3] has been administered in the primary study NCT00294047.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to enrolment.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A subject previously enrolled in the study NCT00294047 and who fulfils either of the following criteria:

  * displayed normal cervical cytology but tested positive for oncogenic HPV infection at her concluding NCT00294047 study visit
  * was pregnant so that no cervical sample could be collected at her concluding NCT00294047 study visit

Exclusion Criteria:

* A subject who at the NCT00294047 concluding study visit displayed normal cervical cytology and who was negative for oncogenic HPV infection at that visit.
* A subject who at the NCT00294047 concluding study visit had a cervical lesion at that visit or who had a cervical lesion that required treatment at her NCT00294047 exit colposcopy.
* A subject for whom the cervical cytology results from the concluding NCT00294047 study visit were unavailable for reasons other than pregnancy.

Min Age: 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (3):
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Wenatchee, Washington
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- Portugal (4):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Setúbal
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Singapore, Singapore
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=113617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by multiple investigators at 20 centres in Canada, Netherlands, Portugal, Russian Federation, Singapore, United Kingdom and the United States.
Pre-assignment Details: Although 34 subjects were enrolled in the study, 2 were excluded following eligibility criteria, leading to 32 subjects who started the study.
Period: Overall Study
Arm/Group | HPV-062 Study Subjects Group
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 28
  Asian - South East Asian Heritage | 2
  African Heritage / African American | 1
  American Indian or Alaskan Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Positive Oncogenic HPV DNA Results by Hybrid Capture II Test (HCII) at Month 12
Description: Subjects with 2 positive oncogenic HPV DNA tests or 1 cervical cytology reading ≥ASC-US (atypical squamous cells of undetermined significance) positive for oncogenic HPV DNA or 1 cervical cytology reading ≥LSIL (low grade squamous intraepithelial lesion) were referred for colposcopy evaluation according to the clinical management algorithm.
Time Frame: At Month 12 [12 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: The analysis was performed on the Total HPV-062 cohort, which included subjects from HPV-015 study who displayed normal cervical cytology, but tested positive for oncogenic HPV infection at their concluding HPV-015 study visit, or who were pregnant at their concluding study visit, and for whom data were available at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 13
Participants | 2

2. Primary Outcome: Number of Subjects Reporting Positive Oncogenic HPV DNA Results by Hybrid Capture II Test (HCII) at Month 24
Description: as for outcome 1
Time Frame: At Month 24 [24 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: The analysis was performed on the Total HPV-062 cohort, which included subjects from HPV-015 study who displayed normal cervical cytology, but tested positive for oncogenic HPV infection at their concluding HPV-015 study visit, or who were pregnant at their concluding study visit, and for whom data were available at Month 24.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 12
Participants | 3

3. Primary Outcome: Number of Subjects Reporting Positive Oncogenic HPV DNA Results by Hybrid Capture II Test (HCII) at Month 36
Description: as for outcome 1
Time Frame: At Month 36 [36 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: The analysis was performed on the Total HPV-062 cohort, which included subjects from HPV-015 study who displayed normal cervical cytology, but tested positive for oncogenic HPV infection at their concluding HPV-015 study visit, or who were pregnant at their concluding study visit, and for whom data were available at Month 36.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 9
Participants | 3

4. Primary Outcome: Number of Subjects Reporting Positive Oncogenic HPV DNA Results by Hybrid Capture II Test (HCII) at Month 48
Description: as for outcome 1
Time Frame: At Month 48 [48 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: The analysis was performed on the Total HPV-062 cohort, which included subjects from HPV-015 study who displayed normal cervical cytology, but tested positive for oncogenic HPV infection at their concluding HPV-015 study visit, or who were pregnant at their concluding study visit, and for whom data were available at Month 48.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 6
Participants | 1

5. Primary Outcome: Number of Subjects With Any Cytological Abnormalities in Cervical Samples by ThinPrep PapTest at Month 12
Description: Cytological abnormalities = atypical squamous cells of undetermined significance (ASC-US).
  Cervical cytology was performed using the ThinPrep PapTest by Quest Diagnostics, or another GSK designated laboratory. Cervical cells for ThinPrep cytology were collected using the sampling device provided and rinsed into a collection vial containing PreservCyt medium.
Time Frame: At Month 12 [12 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 15
Participants
  Normal | 11
  ASC-US | 2
  LSIL | 2

6. Primary Outcome: Number of Subjects With Any Cytological Abnormalities in Cervical Samples by ThinPrep PapTest at Month 24
Description: as for outcome 5
Time Frame: At Month 24 [24 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 12
Participants
  Normal | 11
  ASC-US | 1
  LSIL | 0

7. Primary Outcome: Number of Subjects With Any Cytological Abnormalities in Cervical Samples by ThinPrep PapTest at Month 36
Description: as for outcome 5
Time Frame: At Month 36 [36 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 9
Participants
  Normal | 8
  ASC-US | 1
  LSIL | 0

8. Primary Outcome: Number of Subjects With Any Cytological Abnormalities in Cervical Samples by ThinPrep PapTest at Month 48
Description: as for outcome 5
Time Frame: At Month 48 [48 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 6
Participants
  Normal | 6
  ASC-US | 0
  LSIL | 0

9. Primary Outcome: Number of Subjects With Referral to Colposcopy at Month 12
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: At Month 12 [12 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 15
Participants
  Colposcopy referral: Yes | 4
  Colposcopy referral: No | 11
  Colposcopy performed: Yes | 4
  Colposcopy performed: No | 11
  Algorithm respected: number analyzed (Participants) | 4
  Algorithm respected: Yes | 4
  Algorithm respected: No | 0
  Lesion: number analyzed (Participants) | 4
  Lesion: Yes | 1
  Lesion: No | 3

10. Primary Outcome: Number of Subjects With Referral to Colposcopy at Month 24
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: At Month 24 [24 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 12
Participants
  Colposcopy referral: Yes | 1
  Colposcopy referral: No | 11
  Colposcopy performed: Yes | 1
  Colposcopy performed: No | 11
  Algorithm respected: number analyzed (Participants) | 1
  Algorithm respected: Yes | 1
  Algorithm respected: No | 0
  Lesion: number analyzed (Participants) | 1
  Lesion: Yes | 0
  Lesion: No | 1

11. Primary Outcome: Number of Subjects With Referral to Colposcopy at Month 36
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: At Month 36 [36 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 9
Participants
  Colposcopy referral: Yes | 3
  Colposcopy referral: No | 6
  Colposcopy performed: Yes | 3
  Colposcopy performed: No | 6
  Algorithm respected: number analyzed (Participants) | 3
  Algorithm respected: Yes | 3
  Algorithm respected: No | 0
  Lesion: number analyzed (Participants) | 3
  Lesion: Yes | 0
  Lesion: No | 3

12. Primary Outcome: Number of Subjects With Referral to Colposcopy at Month 48
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: At Month 48 [48 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 6
Participants
  Colposcopy referral: Yes | 1
  Colposcopy referral: No | 5
  Colposcopy performed: Yes | 2
  Colposcopy performed: No | 4
  Algorithm respected: number analyzed (Participants) | 2
  Algorithm respected: Yes | 1
  Algorithm respected: No | 1
  Lesion: number analyzed (Participants) | 2
  Lesion: Yes | 0
  Lesion: No | 2

13. Primary Outcome: Number of Subjects With Referral to Treatment at Month 12
Description: If a high-grade lesion was observed, the subject was referred to treatment according to local medical practice. Any further management following local cervical therapy for cervical lesions was handled according to local medical practice within the local health care system. After treatment, the subject's participation in the study ended.
Time Frame: At Month 12 [12 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 4
Participants
  Treatment referral: Yes | 0
  Treatment referral: No | 4
  Treatment done: Yes | 0
  Treatment done: No | 4

14. Primary Outcome: Number of Subjects With Referral to Treatment at Month 24
Description: as for outcome 13
Time Frame: At Month 24 [24 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 1
Participants
  Treatment referral: Yes | 0
  Treatment referral: No | 1
  Treatment done: Yes | 0
  Treatment done: No | 1

15. Primary Outcome: Number of Subjects With Referral to Treatment at Month 36
Description: as for outcome 13
Time Frame: At Month 36 [36 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 3
Participants
  Treatment referral: Yes | 1
  Treatment referral: No | 2
  Treatment done: Yes | 1
  Treatment done: No | 2
  Loop excision of cervix: number analyzed (Participants) | 1
  Loop excision of cervix: Yes | 1
  Loop excision of cervix: No | 0
  Loop cone of cervix: number analyzed (Participants) | 1
  Loop cone of cervix: Yes | 0
  Loop cone of cervix: No | 1
  Cold knife cone of cervix: number analyzed (Participants) | 1
  Cold knife cone of cervix: Yes | 0
  Cold knife cone of cervix: No | 1
  Laser excision cone of cervix: number analyzed (Participants) | 1
  Laser excision cone of cervix: Yes | 0
  Laser excision cone of cervix: No | 1
  Other: number analyzed (Participants) | 1
  Other: Yes | 0
  Other: No | 1

16. Primary Outcome: Number of Subjects With Referral to Treatment at Month 48
Description: as for outcome 13
Time Frame: At Month 48 [48 months post concluding HPV-015 visit (Visit 9, Visit 11 or last HPV-015 study visit)]
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-062 Study Subjects Group
Number analyzed (Participants) | 2
Participants
  Treatment referral: Yes | 0
  Treatment referral: No | 2
  Treatment done: Yes | 0
  Treatment done: No | 2

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs): During the entire study period [from 12 months after concluding HPV-015 (NCT00294047) study visit (Visit 9/Visit 11/Last visit) up to 48 months after concluding HPV-015 (NCT00294047) study visit (Visit 9/Visit 11/Last visit)].
Description: There were no adverse events (AEs) or serious adverse events (SAEs) reported during the entire study period.
Groups:
- HPV-062 Study Subjects Group: HPV-015 (NCT00294047) study subjects who had normal cervical cytology but tested positive for oncogenic HPV infection at their concluding HPV-015 (NCT00294047) study visit or were pregnant so that no cervical sample could be collected at their concluding HPV-015 (NCT00294047) study visit.
Arm/Group | HPV-062 Study Subjects Group
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2010-08-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT01190176/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT01190176/SAP_001.pdf